CLINICAL TRIAL: NCT01684371
Title: The Effects of a Herbal Remedy, Elmore Oil, on Pain and Well-being in Patients With Osteoarthritis: A Double-blind, Placebo-controlled, Randomised Trial.
Brief Title: The Effects of Elmore Oil on Patients With Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Elmore Oil Company Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: EO-01
Record Dates: First submitted 2009-04-22; First posted 2012-09-13 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Degenerative Arthritis; Inflammation
Keywords: Osteoarthritis; Osteoarthritic pain; Arthritic pain; Arthritis; joint inflammation; Arthralgia
MeSH Terms: conditions — Osteoarthritis; Inflammation; Arthritis; Arthralgia | interventions — Tea Tree Oil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blue Dotted Elmore Oil: Patients applied the above oil 3 times daily for four weeks and on the fifth week stopped the application completely for the flush out period before switching to Orange Dotted Elmore Oil
  Interventions: Other: Two oily solutions (Blue Dotted and Orange Dotted Elmore Oils)
- Orange Dotted Elmore Oil: Patients give this oil applied it three times daily on the affected knees for four weeks and on the fifth week, stopped the application totally for the flush out period before switching to the Blue Dotted Elmore Oil.
  Interventions: Other: Two oily solutions (Blue Dotted and Orange Dotted Elmore Oils)

INTERVENTIONS:
Other: Two oily solutions (Blue Dotted and Orange Dotted Elmore Oils) — Thirty participants received Blue Dotted Elmore Oil and another thirty received the Orange dotted Elmore Oil, they applied the oils three times daily on the affected knees for four weeks and stopped usage on the fifth week (flush out period) and on the 6 week, the two group switched to Orange and Blue Elmore Oil respectively. All throughout applications, they filled out their diaries to indicate changes in their mobility, moods, feeling of well being and ability to do their daily work at home or at work every week.
  Other Names: Oily solution in a bottle containing olive oil, tea tree oil, vanilla and eucalyptus.; Another oily solution in a bottle containing olive oil.

SUMMARY:
The treatment of osteoarthritis, a disease that eventually affects the majority of the older population, involves the alleviation of symptoms such as pain and stiffness, and the reduction of inflammation. A double-blind, placebo-controlled, crossover study will be performed to examine the effect of topical application of Elmore Oil, a herbal remedy (containing Eucalyptus oil, Tea tree oil, Olive oil and Vanilla), which has recently been reported to have anti-inflammatory properties, on the symptoms of osteoarthritis.

DETAILED DESCRIPTION:
Sixty patients were randomly selected and approved for the study, 30 patients with even numbers received the blue dotted Elmore oil and 30 patients with odd numbers got the orange dotted Elmore and were advised to apply 3x daily on the affected knees respectively for four weeks. On the fifth week, they stopped application for 7 days as flush out period. Then on the 6th week a cross over was done on the patients - the blue dotted patients, this time received the orange dotted Elmore Oil and vice-versa and did the application three times daily for another 4 weeks. All throughout the usage, they filled out their diaries (noting the degree of pain, feeling of well being (improved sleep, mobility, ability to do their daily activities at home or at work). A pre-application base line laboratory tests were done, after 4 weeks and after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed osteoarthritis based on the criteria developed by the American College of Rheumatology.

Exclusion Criteria:

* Using other forms of topical pain relief.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population from which the cohorts will be selected are from hospital primary care arthritis clinic.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Decrease in joint swelling, pain and stiffness after each treatment period | Every day for 28 days

SECONDARY OUTCOMES:
Detect changes in Full Blood Examination parameters, liver function tests, and kidney function tests, including a CRP and ESR. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Letitia Lucero, MD, Study Director — Veterans Memorial Medical Centre
Locations (1):
- Veterans Memorial Medical Centre, Quezon City, Manila, Philippines

REFERENCES:
- See also: American College of Rheumatology — http://www.rheumatology.org